CLINICAL TRIAL: NCT04812353
Title: Foot and Ankle Arthrodesis or Osteotomy With Io-Fix Type Fixation : a Prospective Study
Brief Title: Foot and Ankle Arthrodesis or Osteotomy With Io-Fix Type Fixation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: S56535
Record Dates: First submitted 2021-03-17; First posted 2021-03-23 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Foot and Ankle Arthrodesis; Foot and Ankle Osteotomy
Keywords: Arthrodesis; Osteotomy; Io-Fix system
MeSH Terms: conditions — Ankylosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Foot and ankle arthrodesis or osteotomy (Other): Patients who underwent a foot- or ankle reconstruction surgery using the Io-Fix system
  Interventions: Other: Follow-up of Io-Fix type fixation

INTERVENTIONS:
Other: Follow-up of Io-Fix type fixation — Follow-up of patients who underwent a foot- or ankle reconstruction surgery using the Io-Fix system

SUMMARY:
The recovery of foot and ankle arthrodesis and osteotomy is still plagued by the problem of delayed consolidation or even pseudo-arthrosis. To date, the foot and ankle unit of UZ Leuven is using a state of the art system, called the Io-Fix system, to optimize the biomechanical stability.

However, the current literature lacks studies assessing and quantifying the advantages of the Io-Fix system. Objective presentations about the use of, and (early) results are currently missing. Therefore, the investigators want to take their responsibility to objectively investigate whether they can confirm and quantify the expected positive results of using the Io-Fix system. Subsequently, the investigators want to search for eventual unexpected problems with Io-Fix.

DETAILED DESCRIPTION:
The recovery of foot and ankle arthrodesis and osteotomy is still plagued by the problem of delayed consolidation or even pseudo-arthrosis. Some known risk factors for delayed consolidation are inherent to the patient and /or cannot be easily corrected by the surgeon: smoking, diabetes mellitus, use of NSAIDS, etc. Many other biological risk factors are well known. The fusion rate is one of these factors. This factor is influenced by the mechanical stability and compression at the level of arthrodesis. The right alignment till the moment of consolidation is an important factor as well.

Currently, two concepts leading to a better fusion rate are under investigation. First, research is done to optimize the local biological factors by using concentrated growth factors. Second, researchers are working towards optimal biomechanical stability and compression by further developing per-operative osteosynthesis material.

Following the optimal biomechanical stability concept, the following innovation was recently released: the Io-Fix system of Extremity Medical L.L.C. (Parsippany , NJ). This state of the art system has clear advantages compared to other systems. Based on the well-expected advantages, the Foot and Ankle unit of UZ Leuven has been using this system since more than one year. The initial subjective results with Io-Fix are strongly positive.

However, the current literature lacks studies assessing and quantifying the advantages of the Io-Fix system. Objective presentations about the use of, and (early) results are currently missing. Therefore, the investigators want to take their responsibility to objectively investigate whether they can confirm and quantify the expected positive results of using the Io-Fix system. Subsequently, the investigators want to search for eventual unexpected problems with Io-Fix.

However, the investigators believe that a larger study groups within a prospective framework with a longer follow-up is mandatory.

ELIGIBILITY:
Inclusion Criteria:

* Being routinely scheduled for a reconstructive surgical procedure for the following indications or involving the following type of procedure

  1. Any reconstructive procedure for Pes Planus, Pes Plano-valgus, or Posterior Tibial Tendon Dysfunction
  2. Tibio-talar arthrodesis or prosthesis
  3. Sub-talar -and/or (partial) Chopart - and/or Triple arthrodesis
  4. Pantalar arthrodesis with or without inclusion of the Chopart joint

     Exclusion Criteria:
* Age under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Radiological and clinical evaluation | within a period of 1 year
  Radiological and clinical evaluation will be combined to determine the fusion rate within a measured time span

SECONDARY OUTCOMES:
Short Form 36 Health Survey Questionnaire (SF-36) | within a period of 1 year
  To capture patients' perceptions of their own health and well-being
American Orthopedic Foot and Ankle Score (AOFAS) | within a period of 1 year
  To measure the outcome of treatment in patients who sustained a complex ankle or hindfoot injury

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided